CLINICAL TRIAL: NCT01464567
Title: Comparison Between Spontaneous Breathing Trials Through Pressure-Support Ventilation or "T" Tube in the Weaning of Mechanical Ventilation in Patients With Chronic Obstructive Pulmonary Disease: A Randomized Controlled Trial
Brief Title: Spontaneous Breathing Trials Using Pressure-Support or T-Tube in Chronic Obstructive Pulmonary Disease Patients Weaning Mechanical Ventilation
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Hospital Nossa Senhora da Conceicao (Other)
Responsible Party: Principal Investigator, Jose Augusto Santos Pellegrini, Principal Investigator, Hospital Nossa Senhora da Conceicao
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: TVEDPOC-001
Record Dates: First submitted 2011-10-24; First posted 2011-11-03 (Estimated); Last update posted 2016-11-25 (Estimated); Status verified 2016-11

CONDITIONS: Weaning of Mechanical Ventilation; Chronic Obstructive Pulmonary Disease
Keywords: Weaning; Chronic Obstructive Pulmonary Disease; Spontaneous Breathing Trial
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- "T" Tube Spontaneous Breathing Trial (Active Comparator): Spontaneous Breathing Trial wuth "T" Tube for 30 minutes.
  Interventions: Procedure: "T" Tube Spontaneous Breathing Trial
- Pressure Support Ventilation (Experimental): Spontaneous Breathing Trial wuth Ventilation on Pressure-Support mode set at 10cmH2O for 30 minutes
  Interventions: Procedure: Pressure Support Ventilation

INTERVENTIONS:
Procedure: "T" Tube Spontaneous Breathing Trial — "T" Tube ventilation for 30 minutes
  Arms: "T" Tube Spontaneous Breathing Trial
Procedure: Pressure Support Ventilation — Pressure-Support Ventilation for 30 minutes
  Arms: Pressure Support Ventilation

SUMMARY:
Weaning of mechanical ventilation (MV) is an essential part in management of patients with Chronic Obstructive Pulmonary Disease (COPD) when critically ill. The best strategy to be used has not been established.

Objective: To compare the Spontaneous Breathing Trial (SBT) in Pressure Support Ventilation with SBT through "T" tube in weaning of MV in patients with COPD.

Design: Randomized Clinical Trial. Methods: This study will include patients with COPD, admitted to the Intensive Care Unit of Hospital Nossa Senhora da Conceição, undergoing MV for at least 48 hours. When considered by the care team ready for SBT, they will be randomized to one of the following strategies: SBT in Pressure Support or SBT through "T" Tube. The primary endpoint of this study will be the reduction in the days spent on MV. Other outcomes measured will be mortality, extubation and success rate, time to weaning of MV, length of ICU stay and incidence of tracheostomy.

ELIGIBILITY:
Inclusion Criteria:

* COPD patients admitted to our ICU for Acute Respiratory Failure, submitted to Mechanical Ventilation for at least 48 hours
* 18 years or older

Exclusion Criteria:

* Tracheostomy
* Younger than 18 years
* Refuse to give informed consent
* Individuals who are already enrolled in another clinical trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 190 (Actual)
Dates: Start 2012-01; Primary Completion 2016-05 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
Days Spent on Mechanical Ventilation | Participants will be followed for the duration of ICU stay, an expected average of 2 weeks

SECONDARY OUTCOMES:
Mortality | Participants will be followed for the duration of hospital stay, an expected average of 4 weeks
Extubation success rate | Participants will be followed for the duration of ICU stay, an expected average of 4 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Nossa Senhora da Conceição, Porto Alegre, Rio Grande do Sul, Brazil

REFERENCES:
- [Derived] Santos Pellegrini JA, Boniatti MM, Boniatti VC, Zigiotto C, Viana MV, Nedel WL, Marques LDS, Dos Santos MC, de Almeida CB, Dal' Pizzol CP, Ziegelmann PK, Rios Vieira SR. Pressure-support ventilation or T-piece spontaneous breathing trials for patients with chronic obstructive pulmonary disease - A randomized controlled trial. PLoS One. 2018 Aug 23;13(8):e0202404. doi: 10.1371/journal.pone.0202404. eCollection 2018. PMID 30138422